CLINICAL TRIAL: NCT07194031
Title: The Acute Effects of Ankle Exercises on Knee Proprioception and Pain in Individuals With Knee Pain
Brief Title: The Acute Effects of Ankle Exercises on Knee Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Gönül Elpeze, Associated Proffessor, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KNEE PROPRİOCEPTİON
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Knee Pain Chronic
Keywords: Ankle; Exercise; Knee; Pain; Proprioception
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Ankle- Knee Exercises
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee exercise (Active Comparator): Knee flexion-extension
  Interventions: Other: Knee Exercise
- Ankle exercise (Experimental): Ankle plantar flexion with body weight
  Interventions: Other: Ankle Exercise

INTERVENTIONS:
Other: Ankle Exercise — In the literature, studies have evaluated ankle proprioception following interventions applied to the knee. However, no studies report the effects of ankle exercises on knee proprioception
  Other Names: Plantar flexion
  Arms: Ankle exercise
Other: Knee Exercise — The literature emphasizes that long-term and multidirectional exercise programs provide proprioceptive improvements
  Other Names: Knee flexion-extension
  Arms: Knee exercise

SUMMARY:
The goal of this randomized research study is to investigate the acute effects of ankle exercises on improving knee proprioception and pain in individuals with knee pain, aged 18-70, who receive intervention-based ankle and knee exercises to treat their knee pain. The main question it aims to answer is:

• Does ankle exercise affect knee joint proprioception and pain in individuals with knee pain? Researchers will compare ankle exercise (the intervention) with knee exercise (as part of their regular medical care for knee pain) to determine if ankle exercise is effective in improving knee joint proprioception and reducing pain.

Participants will be asked to do exercises and to let the researchers take their measurements.

ELIGIBILITY:
Inclusion Criteria:

* The participants who have a VAS pain score >5,
* The participants who have experienced knee pain for the last six months or longer,
* The participants who volunteered to participate in the study

Exclusion Criteria:

* Individuals who had undergone knee and ankle surgery within the last year
* Individuals who have a VAS pain score below 5
* Individuals who are experiencing ROM limitations in the knee or ankle
* Individuals who have a neurological pathology in the lower extremity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Knee proprioception | 4 weeks
  Knee flexion- extension position

SECONDARY OUTCOMES:
Knee pain | 4 weeks
  Visual Analogue Scale (VAS); Zero, no pain; 10 worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No